CLINICAL TRIAL: NCT04493190
Title: The Effects of Short-term Scapular Control Training on Motor Control in Overhead Athletes With Shoulder Impingement Syndrome
Brief Title: The Effects of Short-term Scapular Control Training in Overhead Athletes With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM108159F
Record Dates: First submitted 2020-06-29; First posted 2020-07-30 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Impingement Syndrome; Scapular Dyskinesis
Keywords: Corticospinal excitability; Transcranial magnetic stimulation; Motor control training; Scapula-focused exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Scapular control training group (Experimental): Participants in these group will be taught how to correctly movement arm overhead. And they will undergo series of movement tasks with mirror and also receive scapular-focused exercises. The difficulty of the movements protocol will increase weekly.
  Interventions: Procedure: Scapular control training
- General exercise group (Experimental): Participants in this group will receive a general strengthening exercise, focusing on the shoulder muscles. And the load will progressively increase weekly.
  Interventions: Procedure: General exercise
- Healthy subject group (No Intervention): No intervention.

INTERVENTIONS:
Procedure: Scapular control training — Participants in this group will learn how to maintain normal scapular position at first. Then they will progress to moving arm with good scapular control with mirror. Afterward, participants will undergo movements protocol which give different directions of arm movements while keeping scapula in a good alignment. They will also receive scapular-focused exercises. The difficulty of the movement protocol will increase weekly. They will be trained three times per week for 6 weeks with an average duration of 30 min per session.
  Arms: Scapular control training group
Procedure: General exercise — Participants in this group will receive a general shoulder strengthening with theraband or dumbbell. Load will increase weekly. They will be trained three times per week for 6 weeks with an average duration of 30 min per session.
  Arms: General exercise group

SUMMARY:
Subacromial impingement syndrome (SIS) is a common disorder of shoulder joint. SIS has been accounted for 44-65 % of all shoulder pain. It is believed that one important contributing factor is scapular dyskinesis. Patients with SIS demonstrates scapular dyskinesis, including decrease in upward rotation, scapular posterior tilt, and external rotation. Altered muscle activity of scapular muscles may contribute to scapular dyskinesis, such as increase in activity of upper trapezius, and decrease in activity of lower trapezius and serratus anterior. In addition to these changes in neuromuscular control, central nervous system may be re-organized in patients with musculoskeletal disorders. Evidence has been reported that center of gravity of motor mapping changes, corticospinal excitability decreases and inhibition increases in patients with shoulder injuries such as instability, rotator cuff tendinopathy and SIS. These corticospinal changes are believed to be related to chronicity of symptoms and lack of treatment effects.

Previous studies have applied many types of treatments to SIS, such as manipulation, taping, and exercises. However, most studies mainly focused on the outcomes of pain and function, few studies investigated changes in neuromuscular control following treatments. Yet, no study has addressed how corticospinal system changes following treatment in patient with shoulder injuries. Motor skill training, which has been widely used in training healthy subjects or patients with neurological disorders, has been shown to change corticospinal systems, including increasing excitability and decreasing inhibition. To our knowledge, no study has integrated the concepts of motor skill learning into a short-term treatment or investigated the effects of motor skill training on corticospinal systems in patients with SIS. The purposes of the study are to investigate the effects of short-term motor skill training on pain, neuromuscular control, corticospinal system in patients with SIS, and also to investigate whether changes in corticospinal parameters will be related to changes in pain, function and neuromuscular control.

ELIGIBILITY:
Inclusion Criteria (patients with shoulder impingement) :

1. perform overhead exercise at least 4 hours a week
2. present type I or II scapular dyskinesis at rest or moving
3. pain at least two weeks
4. 3 of 6 impingement test present positive

   * Neer's impingement test: arm abduction overhead with shoulder internal rotation and thumb downward. If feel pain, then positive.
   * Hawkins-Kennedy impingement Test: arm lift to horizontal plane, elbow flexion to 90 degree. Tester put force on forearm toward shoulder internal rotation. If feel pain, then positive.
   * Empty can test: shoulder abduction with thumb down, then give a resistive force toward up. If feel pain, then positive.
   * Resistive shoulder external rotation test: elbow flexion to 90 degrees and do resistive shoulder rotation. If feel pain, then positive.
   * Rotator cuff tenderness test: tester put pressure on rotator cuff. If feel pain, then positive.
   * Painful arc: perform arm elevation. If feel pain during movement, then positive.

Inclusion Criteria (healthy people) :

1. perform overhead exercise at least 4 hours a week
2. no any symptoms or injuries on shoulder and neck

Exclusion Criteria:

1. Have a history of dislocation, fracture, or surgery of upper extremity
2. A history of direct contact injury to the neck or upper extremities within the past 12 months
3. A concussion within the past 12 months or a history of three or more concussions
4. Brain injury and neurological impairment
5. History of frequent headache or dizziness
6. Contraindications to the use of transcranial magnetic stimulation (TMS), assessed with a safety screening questionnaire, including pregnancy, history of seizure, epilepsy and syncope, having cochlear implant, having medal implant and taking anti-depressant medication.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Change in neurophysiological measures - Active motor threshold | Change from baseline AMT at 6 weeks
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Change in neurophysiological measures - Motor evoked potential | Change from baseline MEP at 6 weeks
  Motor evoked potential (MEP) will be described with millivolt (mV) at different points and with different stimulus intensity
Change in neurophysiological measures - Cortical silent period | Change from baseline CSP at 6 weeks
  Cortical silent period (CSP) will be measured with millisecond (ms).
Change in neurophysiological measures - Short interval cortical inhibition and short interval cortical facilitation | Change from baseline SICI and SICF at 6 weeks
  Short interval cortical inhibition (SICI) and short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses
Change in shoulder pain | Change from baseline pain at 6 weeks
  Pain will be measured with a numerical rating scale (0-10). Zero indicates the absence of pain, while 10 represents the most intense pain possible. No unit.
Change in shoulder function | Change from baseline function at 6 weeks and 3 months
  Function will be measured questionnaire, Flexilevel Scale of Shoulder Function (FLEX-SF). There are 15 questions on each difficulty version. Zero indicates the most difficulty, while 3 means the least difficulty.
Long-term change in shoulder pain | Change from baseline pain at 3 months
  Pain will be measured with a numerical rating scale (0-10). Zero indicates the absence of pain, while 10 represents the most intense pain possible. No unit.
Long-term change in shoulder function | Change from baseline pain at 3 months
  Function will be measured questionnaire, FLEX-SF. There are 15 questions on each

SECONDARY OUTCOMES:
Scapular kinematics | Change from baseline scapular kinematics at 6 weeks
  Including anterior/posterior tilt, upward/downward rotation, and internal/external rotation in scapula plan elevation at 30°, 60°, 90°, and 120°, will be calculated and will be described with degree (°).
Scapular muscle activation | Change from baseline muscle activation at 6 weeks
  The root mean square of electromyography (EMG) data of the upper trapezius, lower trapezius, and serratus anterior will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated over three 30° increments of motion during arm elevation from 30° to 120°, including 30° - 60°, 60° - 90°, and 90° - 120°

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan